CLINICAL TRIAL: NCT00773812
Title: Neuronal Nicotinic Receptor Modulation in the Treatment of Autism: A Pilot Trial of Mecamylamine
Brief Title: Placebo-Controlled Pilot Trial of Mecamylamine for Treatment of Autism Spectrum Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, L. Eugene Arnold, Interim Director of Nisonger Center, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007H0096
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Autistic Disorder; Pervasive Developmental Disorder
Keywords: Autistic Disorder; Autism; Mecamylamine; Pervasive Developmental Disorder-Not Otherwise Specified
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive | interventions — Mecamylamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Mecamylamine (Experimental): There will be 12 children in this arm. These children will receive the active medication (mecamylamine).
  Interventions: Drug: mecamylamine
- Placebo (Placebo Comparator): There will be 8 children in this arm. These children will receive placebo instead of the active medication.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mecamylamine — The dosage is titrated at 6 weeks of .5mg, 2 weeks of 2.5 mg, and 6 weeks of 5.0 mg. One pill is taken once daily.
  Other Names: Inversine
  Arms: Active Mecamylamine
Drug: placebo — One pill is taken once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and efficacy of mecamylamine for the core symptoms of autism.

DETAILED DESCRIPTION:
This is a placebo-controlled pilot clinical trial of a nicotinic agent based on evidence that a disturbance occurs in nicotinic cholinergic transmission in the brain of autistic children. This pharmacotherapeutic trial will be conducted as a direct result of findings of a nicotinic receptor abnormality in autopsied brain tissue from individuals who suffered from autism. A pharmacological agent, mecamylamine, with specificity for the nicotinic receptors implicated in autism, will be tested in children with autism spectrum disorder. Twenty children who meet inclusion/exclusion criteria will be randomized in a 2:3 ratio to 14 weeks of either matched placebo (n=8) or mecamylamine (n=12). Children randomized to placebo who do not respond will be given the opportunity to enroll in a ten week open label extension.

The trial has been completed and published in J. of Child & Adolescent Psychopharmacology.

ELIGIBILITY:
Inclusion Criteria:

* Autistic Disorder or Pervasive Developmental Disorder-Not Otherwise Specified
* Age 4-12
* General good health
* IQ of >=36 or mental age of >=18 months
* Parent/caregiver willingness to accompany child to clinic and monitor for side effects

Exclusion Criteria:

* Unstable Seizure Disorder
* Psychoactive medication in the process of adjustment
* Antipsychotic medication in previous 3 months before baseline
* Systemic corticoids (inhalers allowed)
* Planned beginning of major behavioral intervention in 3 months of study or the 2 months prior to the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary measure will be a global composite derived by calculating the z scores on each measure other than CGI from published norms (or from the baseline descriptives, then averaging the z scores of the various outcome measures for each individual. | Baseline, weeks 2, 4, 6, 8, 10,12, and 14.

SECONDARY OUTCOMES:
OSU Autism Rating Scale-DSM-IV | Baseline, week 6, 8, and 14.
Repetitive Behavior Questionnaire | Baseline, week 2, 4, 6, 8, 10, 12, and 14
Aberrant Behavior Checklist | Baseline, week 2, 4, 6, 8, 10, 12, and 14.
Ohio Autism Clinical Impressions Scale | Baseline, weeks 1, 2, 4, 6, 7, 8, 9, 10, 12, and 14.
Social Responsiveness Scale | Baseline, weeks 2, 4, 6, 8, 10, 12, and 14.
Expressive Vocabulary test-Second Edition | Baseline and week 14
Adverse Experience checklist and AE log | Baseline, weeks 1, 2, 4, 6, 7, 8, 9, 10, 12, and 14.
Cognitive Battery | baseline, weeks 6, 8, and 14

CONTACTS AND LOCATIONS:
Overall Officials: L E Arnold, M.D., Principal Investigator — Ohio State University
Locations (1):
- Nisonger Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Arnold LE, Aman MG, Hollway J, Hurt E, Bates B, Li X, Farmer C, Anand R, Thompson S, Ramadan Y, Williams C. Placebo-controlled pilot trial of mecamylamine for treatment of autism spectrum disorders. J Child Adolesc Psychopharmacol. 2012 Jun;22(3):198-205. doi: 10.1089/cap.2011.0056. Epub 2012 Apr 26. PMID 22537359
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711